CLINICAL TRIAL: NCT05022264
Title: Remote Investigation and Assessment of Vital Signs
Acronym: RIA-VS
Status: Recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: U1111-1261-8273
Record Dates: First submitted 2021-07-29; First posted 2021-08-26 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Blood Pressure; Pulse Rate; Respiratory Rate; Oxygen Saturation; Body Temperature

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: All participants will have their vital signs measured with conventional techniques as well as with the new experimental medical device (labelled RIA-VS)
  Interventions: Diagnostic Test: RIA-VS

INTERVENTIONS:
Diagnostic Test: RIA-VS — Measuring vital signs with a new contactless camera technique
  Other Names: Remote Investigation and Assessment of Vital Signs

SUMMARY:
The vital signs (pulse, systolic and diastolic blood pressure, respiratory rate, oxygen saturation and body temperature) are critical in assessing the severity and prognosis of infections. The devices used today for measuring the vital signs have to be in physical contact with the patients. There is an apparent risk of transferring infections from one patient to the next (or to healthcare professionals). Accurately obtaining vital signs is also important when managing other categories of patients where it may be relevant to obtain some of the vital signs such as pulse and blood pressure.

This project aims to evaluate a new camera-based system for contactless measurement of vital signs.

DETAILED DESCRIPTION:
STUDY DESIGN:

A method comparison design with three work packages (WP):

WP1: Focus on estimating validity and reliability of the new study device to measure body temperature.

WP2: Focus on estimating validity and reliability of the new study device to measure all vital signs except body temperature (pulse, systolic and diastolic blood pressure, respiratory rate and oxygen saturation).

WP3: Focus on estimating if there is any difference in the validity and reliability of the new study device to measure all vital signs (except body temperature) in subjects with Fitzpatrick skin type 5-6 as compared with those of skin type 1-4.

STUDY POPULATION:

WP1: Patients aged ≥18 years admitted to or attending a hospital clinic. WP2: Patients aged ≥18 year attending primary health care or patients being admitted to a hospital clinic.

WP3: Individuals aged ≥18 years attending primary health care.

ELIGIBILITY:
Inclusion Criteria:

The same subject can't be enrolled more than once with the exception that subjects in WP1 may also be recruited to WP2.

WP1+WP2:

1. The patient is attending primary or secondary health care.
2. The subject has provided informed consent.
3. Age ≥18 years.
4. Fluent in Swedish, English, Somali or Arabic (we will translate the patient information and ensure an interpreter can be present for translating questions).
5. The patient is willing and able to give informed consent ".
6. The investigator determines that the new study device, and the reference methods, can be used as intended with adequate safety.
7. The delay in the management of each patient introduced by this study is approximately 15-20 minutes. Patients deemed being in such a severe medical condition that 15-20 minutes of delay is deemed detrimental will not be included.

WP3:

1. Patients attending primary health care.
2. The subject has provided informed consent.
3. Age ≥18 years.
4. Fluent in Swedish, English, Somali or Arabic (we will translate the patient information and ensure an interpreter can be present for translating questions).
5. The patient is willing and able to give informed consent .
6. The investigator determines that the new study device, and the reference methods, can be used as intended with adequate safety.
7. The delay in the management of each patient introduced by this study is approximately 15-20 minutes. Patients deemed being in such a severe medical condition that 15-20 minutes of delay is deemed detrimental will not be included.

Exclusion Criteria:

Subjects are free to withdraw from the study at any point. Subjects will also be withdrawn from the study in case of unexpected depressed level of consciousness from inclusion up until all investigations are completed (during approximately 15-20 minutes). Any reduction in consciousness will incur that the subject is withdrawn.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be consecutive patients attending one of the clinics participating in the study. They will be asked for participation irrespective f reason for attending the clinic. Hence, this study does not focus on any specific medical condition. Participating clinics are one one hospital department for infectious diseases and four clinics for family medicine (general practice / primary health care centers)
Sampling Method: Non-Probability Sample
Enrollment: 860 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Agreement between conventional techniques and the new RIA-VS device | The time delay between the measurements using conventional techniques and the new RIA-VS device will be approximately 5 minutes
  Estimate the agreement between vital signs estimated with the new RIA-VS study device and vital signs estimated using traditional techniques (the criterion validity). Vital signs in this context are heart rate (pulse), respiratory rate, oxygen saturation (SpO2), systolic as well as diastolic blood pressure, and body temperature. For each vital sign the following statistics will be calculated to answer the outcome measure:
  a) Validity of the new method: The gold standard will be the mean between the two reference methods. The first measurement of the new RIA-VS device will be the new method compared with the gold standard using a Bland-Altman plot. We will also produce simple scatter plots comparing the gold standard with the new RIA-VS device for illustration.

SECONDARY OUTCOMES:
Estimate test-retest reliability of the new RIA-VS device | The time delay between the measurements using conventional techniques and the new RIA-VS device will be approximately 5 minutes
  Estimate the new RIA-VS study device test-retest reliability and to compare this with the test-retest reliability of the reference method. Vital signs in this context are heart rate (pulse), respiratory rate, oxygen saturation (SpO2), systolic as well as diastolic blood pressure, and body temperature. For each vital sign the following statistics will be calculated to answer the outcome measure:
  1. Test-retest reliability of the new RIA-VS method: The difference between the two tests will be plotted on the Y-axis and the mean value of the two estimates of the new RIA-VS device on the x-axis in a modified Bland-Altman plot.
  2. Comparison of the random variability: The variance of the difference between the two measures using the reference method will be compared with the variance from the difference between the two RIA-VS estimates. This enables comparing the random variability of both the reference method as well as the new RIA-VS device.
Evaluate the influence of different skin types on the validity of the new RIA-VS study device | The time delay between the measurements using conventional techniques and the new RIA-VS device will be approximately 5 minutes
  Investigate if different Fitzpatrick skin types influences the validity of the new RIA-VS study device. We will use the definition of skin types as described in: Fitzpatrick TB. The validity and practicality of sun-reactive skin types I through VI. Arch Dermatol. 1988;124(6):869-71).
  The statistics described in the primary outcome measure and the first secondary outcome measure (test-retest reliability) will be made separately for patients with Fitzpatrick skin color type 0-4 as well as type 5-6 to see if skin color influences readings with the new RIA-VS device.

CONTACTS AND LOCATIONS:
Overall Officials: Ronny Gunnarsson, MD PhD, Principal Investigator — School of Public Health and Community Medicine, Gothengurg University, Sweden
Locations (1):
- Hälsobrunnen Vårdcentral, Ulricehamn, Sweden

IPD SHARING:
Plan to Share IPD: Yes
A deidentified raw data file will be publicly available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Raw data will be made available upon acceptance of final manuscript for publication
Access Criteria: Publicly available to anyone